CLINICAL TRIAL: NCT02673372
Title: Low-Dose Ketamine Versus Morphine for Moderate to Severe Pain in the Emergency Department Geriatric Population: A Prospective, Randomized, Double-Blind Study.
Brief Title: Geriatric Ketamine for Pain Management Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Antonios Likourezos (Other)
Responsible Party: Sponsor-Investigator, Antonios Likourezos, Research Manager, Maimonides Medical Center
Organization: Maimonides Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2015-10-14; 2015-10-14 (Other: Maimonides Medical Center)
Record Dates: First submitted 2016-02-01; First posted 2016-02-03 (Estimated); Results first posted 2019-05-31 (Actual); Last update posted 2019-05-31 (Actual); Status verified 2019-05

CONDITIONS: Pain
Keywords: Geriatric, Pain, Ketamine, Emergency Medicine
MeSH Terms: conditions — Pain | interventions — Morphine; Ketamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Morphine Group (Active Comparator): intravenous Morphine given at 0.1 mg/kg as intravenous infusion (10 min) with a maximum dose of 10 mg.
  Interventions: Drug: Morphine
- Ketamine Group (Experimental): Ketamine administered in sub-dissociative doses 0.3 mg/kg as a intravenous infusion (10 min)
  Interventions: Drug: Ketamine

INTERVENTIONS:
Drug: Morphine — intravenous Morphine given at 0.1 mg/kg as intravenous infusion (10 min) with a maximum dose of 10 mg. The device is the Care Fusion Alaris PC.
  Arms: Morphine Group
Drug: Ketamine — Ketamine administered in sub-dissociative doses 0.3 mg/kg as a intravenous infusion (10 min). The device is the Care Fusion Alaris PC.
  Arms: Ketamine Group

SUMMARY:
This research project is geared towards geriatric analgesia in the Emergency Department (ED) with a goal of reducing the administration of opioid pain medications to elderly patients, thereby avoiding the commonly occurring, severe side effects associated with such medications, including hypotension, respiratory depression, altered mental status, delirium, as well as nausea/vomiting and constipation.

The primary outcome of the study will be difference in pain score from baseline to 30 minutes post-medication administration.

This project has the potential to change and modify the ED approach to geriatric analgesia by virtue of minimizing the use of opioid administration in elderly patients. T

DETAILED DESCRIPTION:
Elderly patients are making up a greater proportion of the New York State population every year as the nation's overall population continues to age at a rapid pace. Acute and chronic pain conditions are very common in the geriatric population and it is well recognized that pain is undertreated in the elderly. Complicating this important public health problem is that changes in physiology that occur in the elderly, such as cognitive decline and impaired ability of the liver and kidney to metabolize medications, render opioid administration particularly dangerous in the geriatric population. Adverse side effects and increased health care utilization are well known hazards associated with opioid use in the elderly.

Therefore, development of pain management strategies that include non-opioid pain treatment modalities has the potential to have a major impact on the health and well-being of New Yorkers. This study undertakes a novel strategy intended to reduce opioid consumption in the elderly.

This research project will evaluate the analgesic feasibility and safety of short infusion of subdissociative dose of intravenous ketamine compared with short infusion of intravenous morphine for controlling pain in ED patients 65 years of age and older, laying the groundwork for ketamine to become a safe and viable alternative to opioids in managing geriatric pain in the ED. The significance of this project being done at Maimonides Medical center is to lay the foundation to providing safer analgesia in geriatric ED patients and moving towards an eventual goal of an "opioid-free" ED.

Methods:

Study Design:

This is a prospective, randomized, double-blind trial evaluating and comparing analgesic effect of Ketamine administered in sub-dissociative doses 0.3 mg/kg as a intravenous infusion (10 min), and intravenous Morphine given at 0.1 mg/kg as intravenous infusion (10 min) with a maximum dose of 10 mg. in elderly adults (age 65 and older) with pain in the ED.

Study

Protocol:

Patient screening, enrollment, and data collection will be performed by study investigators and the research fellow. ED pharmacy investigators will maintain the randomization list which will be generated prior to commencement of the study, will prepare the medication, and will deliver it to the nurse caring for the study participant in a blinded fashion.

The study will include patients aged 65 and older presenting to the ED with abdominal, flank, back, traumatic chest or musculoskeletal pain of (moderate to very severe pain) five or more on a standard eleven point (0 - 10; with 0 being no pain to 10 very severe pain) numeric rating scale (NRS), and who require opioid analgesia as determined by the treating ED attending physician.

Exclusion criteria will include altered mental status, allergy to morphine or ketamine, weight <40kg or >115kg, unstable vital signs (systolic blood pressure <90 or >200 mmHg, heart rate <50 or >150 beats per minute, non-traumatic chest pain, headache, and respirations <8 or >30 per minute), past medical history of severe renal or hepatic insufficiency, alcohol or drug abuse or psychiatric illness; BMI >40; severe COPD

After patients are evaluated by the treating ED physician and determined to meet eligibility criteria, each patient will be approached by a member of the research team for acquisition of written informed consent and HIPAA authorization. The on-duty ED pharmacist will prepare medications according to the two arms of the study: patients receiving 0.1 mg /kg of morphine ; patients receiving 0.3 mg/kg of ketamine.

The medication will be administered using infusion pump with a 10 minute run time.

Patients a priori will will be randomized to either of the two arms. A list will be generated via SPSS 19.0 from 1 to 90; and SPSS 19.0 will be programmed to randomly assign patients to either of the two arms at 10 patient blocks. Thus, for example in patients 1 to 10; SPSS will randomly assign 5 patients to the Ketamine group and 5 patients to the morphine group and so on for all 90 patients. Therefore, after completion 45 patients will be assigned to the Ketamine group and 45 to the morphine group. Antonios will then e-mail the list to Nicholas Filk and pharmacy department who will have the list and when a patient is enrolled in the study will know which medication to give the patient. Every other investigator and clinician would be blinded to the randomization assignment.

Study investigators will record pain scores, vital signs, and adverse effects at 0, 30, 60, 90, and 120 minutes.

Patients who report a pain NRS of five or greater and request additional pain relief will be given fentanyl 0.5 mcg/kg as a rescue analgesic. All data, including gender, demographics, medical history, and vital signs, will be recorded on data collection sheets and will be entered into and analyzed via SPSS 19.0.

Development of the randomization list, confirmation of written consent acquisition on all participants, and statistical analyses will be conducted by the research manager and statistician, who will be independent of any data collection.

ELIGIBILITY:
Inclusion Criteria:

* ED patients; 65 years of age and older; abdominal, flank, back, traumatic chest, neck or musculoskeletal pain; capacity to give verbal or written consent.

Exclusion Criteria:

* ED patients <65 years old; altered mental status; presenting with headache, non-traumatic chest pain; allergy to morphine or ketamine; weight <40kg or >115kg, unstable vital signs (systolic blood pressure <90 or >180 mmHg; heart rate <5 or >150 beats per minute; and respirations <8 or >30 per minute), and past medical history of severe renal or hepatic insufficiency, alcohol or drug abuse or psychiatric illness; Patients with BMI>40; severe COPD

Ages: 65 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 60 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2018-02 (Actual); Study Completion 2018-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sergey Motov, MD, Principal Investigator — Maimonides Medical Center
Locations (1):
- Maimonides Medical Center, Brooklyn, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gibson SJ. Pain and ageing: a comparison of the pain experience over the adult life span. Prog Pain Res Manage. 2003;24:767-90.
- [Background] Gibson SJ, Farrell M. What is different about pain in older people? Reviews in Analgesia. 2004;8:23-37.
- [Background] Gibson SJ. Older Persons' Pain: what can we learn? Pain Clin Updat. 2006;14:1-4.
- [Background] American Geriatrics Society Panel on the Pharmacological Management of Persistent Pain in Older Persons. Pharmacological management of persistent pain in older persons. Pain Med. 2009 Sep;10(6):1062-83. doi: 10.1111/j.1526-4637.2009.00699.x. Epub 2009 Sep 9. No abstract available. PMID 19744205
- [Background] Leveille SG, Jones RN, Kiely DK, Hausdorff JM, Shmerling RH, Guralnik JM, Kiel DP, Lipsitz LA, Bean JF. Chronic musculoskeletal pain and the occurrence of falls in an older population. JAMA. 2009 Nov 25;302(20):2214-21. doi: 10.1001/jama.2009.1738. PMID 19934422
- [Background] Linnebur SA, O'Connell MB, Wessell AM, McCord AD, Kennedy DH, DeMaagd G, Dent LA, Splinter MY, Biery JC Jr, Chang F, Jackson RC, Miller SL, Sterling T; ACCP Task Force. Pharmacy practice, research, education, and advocacy for older adults. Pharmacotherapy. 2005 Oct;25(10):1396-430. doi: 10.1592/phco.2005.25.10.1396. PMID 16185185
- [Background] Dunn KM, Saunders KW, Rutter CM, Banta-Green CJ, Merrill JO, Sullivan MD, Weisner CM, Silverberg MJ, Campbell CI, Psaty BM, Von Korff M. Opioid prescriptions for chronic pain and overdose: a cohort study. Ann Intern Med. 2010 Jan 19;152(2):85-92. doi: 10.7326/0003-4819-152-2-201001190-00006. PMID 20083827
- [Background] Solomon DH, Rassen JA, Glynn RJ, Lee J, Levin R, Schneeweiss S. The comparative safety of analgesics in older adults with arthritis. Arch Intern Med. 2010 Dec 13;170(22):1968-76. doi: 10.1001/archinternmed.2010.391. PMID 21149752
- [Background] Domino EF. Taming the ketamine tiger. 1965. Anesthesiology. 2010 Sep;113(3):678-84. doi: 10.1097/ALN.0b013e3181ed09a2. PMID 20693870
- [Background] Strigo IA, Duncan GH, Bushnell CM, Boivin M, Wainer I, Rodriguez Rosas EM, Persson J. The effects of racemic ketamine on painful stimulation of skin and viscera in human subjects. Pain. 2005 Feb;113(3):255-264. doi: 10.1016/j.pain.2004.10.023. PMID 15661431
- [Background] Smith DC, Mader TJ, Smithline HA. Low dose intravenous ketamine as an analgesic: a pilot study using an experimental model of acute pain. Am J Emerg Med. 2001 Oct;19(6):531-2. doi: 10.1053/ajem.2001.27152. No abstract available. PMID 11593484
- [Background] Sadove MS, Shulman M, Hatano S, Fevold N. Analgesic effects of ketamine administered in subdissociative doses. Anesth Analg. 1971 May-Jun;50(3):452-7. No abstract available. PMID 5103784
- [Background] Schmid RL, Sandler AN, Katz J. Use and efficacy of low-dose ketamine in the management of acute postoperative pain: a review of current techniques and outcomes. Pain. 1999 Aug;82(2):111-125. doi: 10.1016/S0304-3959(99)00044-5. PMID 10467917
- [Background] Galinski M, Dolveck F, Combes X, Limoges V, Smail N, Pommier V, Templier F, Catineau J, Lapostolle F, Adnet F. Management of severe acute pain in emergency settings: ketamine reduces morphine consumption. Am J Emerg Med. 2007 May;25(4):385-90. doi: 10.1016/j.ajem.2006.11.016. PMID 17499654
- [Background] Jennings PA, Cameron P, Bernard S, Walker T, Jolley D, Fitzgerald M, Masci K. Morphine and ketamine is superior to morphine alone for out-of-hospital trauma analgesia: a randomized controlled trial. Ann Emerg Med. 2012 Jun;59(6):497-503. doi: 10.1016/j.annemergmed.2011.11.012. Epub 2012 Jan 13. PMID 22243959
- [Background] Lester L, Braude DA, Niles C, Crandall CS. Low-dose ketamine for analgesia in the ED: a retrospective case series. Am J Emerg Med. 2010 Sep;28(7):820-7. doi: 10.1016/j.ajem.2009.07.023. Epub 2010 Apr 2. PMID 20837262
- [Background] Ahern TL, Herring AA, Miller S, Frazee BW. Low-Dose Ketamine Infusion for Emergency Department Patients with Severe Pain. Pain Med. 2015 Jul;16(7):1402-9. doi: 10.1111/pme.12705. Epub 2015 Feb 3. PMID 25643741
- [Background] Beaudoin FL, Lin C, Guan W, Merchant RC. Low-dose ketamine improves pain relief in patients receiving intravenous opioids for acute pain in the emergency department: results of a randomized, double-blind, clinical trial. Acad Emerg Med. 2014 Nov;21(11):1193-202. doi: 10.1111/acem.12510. PMID 25377395
- [Background] Motov S, Rockoff B, Cohen V, Pushkar I, Likourezos A, McKay C, Soleyman-Zomalan E, Homel P, Terentiev V, Fromm C. Intravenous Subdissociative-Dose Ketamine Versus Morphine for Analgesia in the Emergency Department: A Randomized Controlled Trial. Ann Emerg Med. 2015 Sep;66(3):222-229.e1. doi: 10.1016/j.annemergmed.2015.03.004. Epub 2015 Mar 26. PMID 25817884
- [Derived] Motov S, Mann S, Drapkin J, Butt M, Likourezos A, Yetter E, Brady J, Rothberger N, Gohel A, Flom P, Mai M, Fromm C, Marshall J. Intravenous subdissociative-dose ketamine versus morphine for acute geriatric pain in the Emergency Department: A randomized controlled trial. Am J Emerg Med. 2019 Feb;37(2):220-227. doi: 10.1016/j.ajem.2018.05.030. Epub 2018 May 16. PMID 29807629

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Morphine Group | Ketamine Group
Started | 30 | 30
Completed | 30 | 30
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Morphine Group | Ketamine Group | Total
Number analyzed (Participants) | 30 | 30 | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 2 | 2 | 4
  >=65 years | 28 | 28 | 56
Age, Continuous [Mean (Standard Deviation); unit: years] | 77.13 (8.51) | 77.27 (8.44) | 77.2 (8.41)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 23 | 46
  Male | 7 | 7 | 14
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 7 | 5 | 12
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 1 | 4
  White | 11 | 21 | 32
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 9 | 3 | 12
Region of Enrollment [Number; unit: participants]
  United States | 30 | 30 | 60

OUTCOME MEASURES:

1. Primary Outcome: Reduction of Pain Score at 30 Minutes
Description: The primary outcome will be the comparative reduction of NRS pain scores between the 2 groups at 30 minutes. The NRS Pain scale ranges from 0 to 10 (0 being no pain at all to 10 being very severe pain; 5 is moderate pain)
Time Frame: 30 minutes
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Morphine Group | Ketamine Group
Number analyzed (Participants) | 30 | 30
score on a scale | 4.4 (3.1) | 4.2 (3.4)

ADVERSE EVENTS:
Time Frame: 30 minutes
Arm/Group | Morphine Group | Ketamine Group
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 2/30 | 2/30
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Morphine Group (N=30) | Ketamine Group (N=30)
Nausea (General disorders) | 2 (2) | 2 (2) — Nausea at 30 minutes

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-10-01): https://cdn.clinicaltrials.gov/large-docs/72/NCT02673372/Prot_SAP_000.pdf